CLINICAL TRIAL: NCT06796816
Title: Bioimpedance Analysis in Perioperative Assessment in Thoracic Surgery
Acronym: BIVA-18
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 945/2018/SPER/IRCCSRE
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Lung Resection; Adenocarcinoma of Lung
Keywords: bioimpedence; lung cancer; sarcopenia
MeSH Terms: conditions — Adenocarcinoma of Lung; Lung Neoplasms; Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients undergoing surgery for removal of adenocarcinoma of the lung (Experimental)
  Interventions: Other: Bioelectrical Impedance Vector Analysis (BIVA)

INTERVENTIONS:
Other: Bioelectrical Impedance Vector Analysis (BIVA) — Bioelectrical Impedance Vector Analysis (BIVA) both in total body mode (Total Body Water) and segmental mode. The device used is the "BIA 101 Anniversary" by Akern. The BIVA exam will be performed in total body and segmental modes.
  For total body mode, the patient should be placed on a non-conductive surface. After cleansing the skin with alcohol or mild soap, 4 electrodes will be placed: 2 on the right hand (metacarpal area) and 2 on the right foot (metatarsal). The cable connected to your instrument will then be connected to the electrodes. After the instrument is switched on, the variables are read and then analysed. For segmental mode, the patient should be placed on a non-conductive surface. After cleansing the skin with alcohol or mild soap, 8 electrodes will be placed: 2 on the right hand (metacarpal area) and 2 on the left hand, 2 on the right foot (metatarsal) and 2 on the left foot.

SUMMARY:
The assessment of surgical and postoperative risks in thoracic surgery is a field of significant interest because the surgical procedure causes substantial changes in the body's homeostasis.

The postoperative course is characterized by considerable clinical variability compared to the preoperative classification, which highlights more homogeneous data among various patient groups. This variability appears to result from individual differences in response to extensive pulmonary resections. Notably, the homogeneity of preoperative data does not correlate with the greater variability observed in the postoperative course.

The application of algorithms derived from BIVA in bioimpedance studies has proven particularly useful for prognostic assessments in oncology, as it can evaluate a patient's hydration status and muscle reserves at the time of diagnosis or the start of clinical/surgical treatment.

Understanding body composition, particularly the quantity and/or quality of muscle mass, is essential for diagnosing sarcopenia.

By passing a low-intensity alternating current (imperceptible to the patient) through the body, BIVA measures provide insights into body water distribution (both intracellular and extracellular), lean mass and skeletal muscle mass. Overall, the test offers a detailed picture of hydration status and skeletal muscle composition.

Another validated tool for assessing sarcopenia, which provides information on both muscle quantity (via cross-sectional area measurements) and muscle quality (via muscle density measurements), is computed tomography (CT). CT imaging is typically performed for diagnostic and staging purposes before surgery in thoracic surgery patients, either alone or in combination with positron emission tomography (PET).

Our study will focus on assessing correlations between clinical, imaging, and bioimpedance data and postoperative outcomes, with particular attention to the incidence of atrial fibrillation (AF), pulmonary atelectasis requiring treatment, and increased pleural drainage production.

Additionally, we will evaluate the relationship between the surgical approach (open surgery vs. video-assisted thoracoscopic surgery, or VATS) and short-term bioimpedance values.

ELIGIBILITY:
Inclusion Criteria:

- Patients undergoing pulmonary resection surgery for primary neoplasm within a one-year timeframe.

Exclusion Criteria:

* Patients with chronic atrial fibrillation (AF).
* Patients who have previously undergone major pulmonary resection.
* Patients with pacemakers or implantable devices, as the use of bioimpedance vector analysis (BIVA) may be contraindicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2019-04-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Body composition | Day 1, day 2 or 3 and day 45 after surgery
  Bioimpedence (total body and segmental)

OTHER OUTCOMES:
Correlation between preoperative body composition and postoperative course, including the possible occurrence of complications in the cardiopulmonary area | Day 1, day 2 or 3 andday 45 after surgery
  Body composition
Correlation between the operating method (open vs VATS) with short-term impedance values | Day 1, day 2 or 3 and day 45 after surgery
  Body composition
Correlation between CT/PET data on sarcopenia collected at the preoperative examination and occurrence of pulmonary atelectasis | Pre e post surgery (staging/re-staging TC, usually performed within 2 months from surgery)
  CT/PET data on sarcopenia will be collected from scans without contrast agents during CT or PET-CT staging, selecting the scan closest to surgery. Parameters measured include cross-sectional area of the pectoral muscle, abdominal muscles (abdominal, psoas, paravertebral) at L3, and thigh root muscles; skeletal muscle index (area/height²) at the pectoral muscle, abdominal muscles at L3, and thigh root; skeletal muscle density (mean HU) at the pectoral muscle, abdominal muscles at L3, and thigh root; intramuscular adipose tissue (IMAT) in these regions; and visceral (VAT) and subcutaneous (SAT) adipose tissue at L3. Data will be analyzed using OsiriX software, selecting slices for each level, setting density windows (-29 to 150 HU for muscle, -30 to -190 HU for adipose tissue), and manually plotting regions of interest (ROI).

CONTACTS AND LOCATIONS:
Locations (1):
- AUSL IRCCS di Reggio Emilia, Reggio Emilia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Belfiore A, Cataldi M, Minichini L, Aiello ML, Trio R, Rossetti G, Guida B. Short-Term Changes in Body Composition and Response to Micronutrient Supplementation After Laparoscopic Sleeve Gastrectomy. Obes Surg. 2015 Dec;25(12):2344-51. doi: 10.1007/s11695-015-1700-0. PMID 25948283
- [Background] Santarelli S, Russo V, Lalle I, De Berardinis B, Navarin S, Magrini L, Piccoli A, Codognotto M, Castello LM, Avanzi GC, Villacorta H, Precht BLC, de Araujo Porto PB, Villacorta AS, Di Somma S; Great Network. Usefulness of combining admission brain natriuretic peptide (BNP) plus hospital discharge bioelectrical impedance vector analysis (BIVA) in predicting 90 days cardiovascular mortality in patients with acute heart failure. Intern Emerg Med. 2017 Jun;12(4):445-451. doi: 10.1007/s11739-016-1581-9. Epub 2016 Dec 16. PMID 27987064
- [Background] Cardoso ICR, Aredes MA, Chaves GV. Applicability of the direct parameters of bioelectrical impedance in assessing nutritional status and surgical complications of women with gynecological cancer. Eur J Clin Nutr. 2017 Nov;71(11):1278-1284. doi: 10.1038/ejcn.2017.115. Epub 2017 Aug 9. PMID 28792014